CLINICAL TRIAL: NCT02107430
Title: Randomized, Open-label, Parallel-group, Multi-centre Phase II Clinical Trial of Active Cellular Immunotherapy With Preparation DCVAC/PCa in Patients With Localized High-risk Prostate Cancer After Primary Radiotherapy
Brief Title: Phase II Study of DCVAC/PCa After Primary Radiotherapy for Patients With High Risk Localized Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SOTIO a.s. (Industry)
Responsible Party: Sponsor
Organization: Sotio Biotech Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP004; 2011-004967-65 (EudraCT Number)
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-09

CONDITIONS: Prostate Cancer
Keywords: Immunotherapy; Prostate Cancer; Biological, Vaccine
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DCVAC/PCa arm post radiotherapy (Experimental): Dendritic Cells DCVAC/PCa Experimental therapy post radiotherapy
  Interventions: Biological: Dendritic Cells DCVAC/PCa
- Standard radiotherapy (Active Comparator): Standard care
  Interventions: Biological: Dendritic Cells DCVAC/PCa; Radiation: Standard radiotherapy

INTERVENTIONS:
Biological: Dendritic Cells DCVAC/PCa — DCVAC/PCa arm post radiotherapy
Radiation: Standard radiotherapy — radiotherapy
  Arms: Standard radiotherapy

SUMMARY:
The purpose of this study is to determine whether DCVAC/PCa added after radical primary prostatectomy can improve PSA progression times within 5 years for patients with high risk localized Prostate Cancer.

DETAILED DESCRIPTION:
Treatment post radical primary prostatectomy Treatment post standard radiotherapy

ELIGIBILITY:
Inclusion Criteria:

* Male 18 years and older
* Histologically confirmed localized prostate cancer of high risk or very high risk fulfilling at least one of the following: T3-T4 stage or Gleason Score 8-10 or PSA level above 20 ng/ml
* Indication for prostate cancer radical radiotherapy
* Neo-adjuvant androgen androgen-deprivation therapy due to prostate cancer using Luteinizing-hormone-releasing hormone (LHRH) analogues ongoing for at least two months and not longer than 12 months prior randomization
* Eastern Cooperative Oncology Group (ECOG) 0-2

Exclusion Criteria:

* Primary surgical treatment of prostate cancer
* Prior or ongoing chemotherapy for prostate cancer
* Participation in other clinical study or administration of other evaluated drug within 30 day prior screening
* Unresolved lasting obstruction of urinary system
* Other uncontrolled inter-current illness
* Treatment with immunotherapy against Prostate Cancer
* Clinically significant cardiovascular disease
* History of primary immunodeficiency
* Active autoimmune disease requiring treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-03; Primary Completion 2013-09 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Number of Prostate Specific Antigen (PSA) failures in 5 years | Enrollment up to 260 weeks
  PSA failure per Phoenix criteria of increase of 2ng/mL over nadir

SECONDARY OUTCOMES:
Proportion of Patients without use of salvage therapy within 5 years | Enrollment up to 260 weeks
  Calculation of the proportion of patients without use of salvage therapy within 5 years
Frequency of Adverse Events | enrollment up to 260 weeks
  Safety profile as defined by the nature, incidence, duration, severity and outcome of adverse events
Proportion of Patients without Objective disease progression within 5 years | Enrollment up to 260 weeks
  Proportion of patients who do not have a >2ng/mL elevation in PSA or require salvage therapy

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Scheiner, Study Director — Sotio Biotech Inc.
Locations (6):
- Czechia (6):
  - Nemocnice Jihlava,Urologické oddělení,, Jihlava
  - Fakultní nemocnice Olomouc, Olomouc
  - FN Ostrava, Onkologická klinika, Ostrava
  - FNKV Klinika radiologie a onkologie, Prague
  - FN Motol, Prague
  - Nemocnice Na Bulovce, Prague

IPD SHARING:
Plan to Share IPD: Yes
Clinical trial results will be reported as required by European legislation in clinicaltrialsregister.eu.
Time Frame: Data will be available 12 months after study completion.
Access Criteria: No specific access criteria are required
URL: https://www.clinicaltrialsregister.eu/ctr-search/search?query=SP004